CLINICAL TRIAL: NCT01040000
Title: A Phase 1/2 Therapeutic, Open Label, Multi-Center Clinical Trial of NPC-1C, a Chimeric Monoclonal Antibody, in Adults With Recurrent, Locally Advanced Unresectable or Metastatic Pancreatic and Colorectal Cancer After Standard Therapy
Brief Title: QUILT-3.019: Phase 2 Study of NPC-1C Chimeric Monoclonal Antibody to Treat Pancreatic and Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precision Biologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neogenix 0901
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Pancreatic Cancer; Metastatic Colorectal Cancer
Keywords: NPC-1C; Monoclonal antibody; Pancreatic Cancer; Adenocarcinoma of the pancreas; Ductal carcinoma of the pancreas; Duct cell carcinomas, pancreas; Carcinomas, pancreas duct cell; Pancreas duct cell carcinoma; Pancreatic duct cell carcinoma; Adenocarcinoma of the colon; Adenocarcinoma of the rectum; Colorectal cancer; Colorectal tumor; Colorectal neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Pancreatic Ductal; Colonic Neoplasms; Rectal Neoplasms | interventions — ensituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPC-1C/NEO-102 (Experimental)
  Interventions: Drug: NPC-1C/NEO-102

INTERVENTIONS:
Drug: NPC-1C/NEO-102 — Subjects will receive NPC-1C at a dose of 3.0 mg/kg. NPC-1C will be given intravenously (by vein) over approximately 1-6 hours, once every 2 weeks for 4 doses per course. Courses will be repeated in the absence of disease progression or unacceptable toxicity.
  Other Names: Ensituximab

SUMMARY:
The purpose of the phase 2 component of this study is to determine if giving the immune molecule NPC-1C to individuals who have cancer of the pancreas or gastrointestinal tract (colon or rectum) which has not responded to standard treatments can shrink or halt the growth of cancer, and to obtain additional data to study its effect on the immune system. Safety data will also be accumulated and evaluated during this study. NPC-1C is a monoclonal antibody that recognizes a specific tumor target on certain cancers. In laboratory studies, the antibody killed tumor cells in some colon and pancreatic cancers that express the NPC-1C antigen by a process called "antibody-dependent cell cytotoxicity" or ADCC.

DETAILED DESCRIPTION:
The limitations of many current therapeutic products for pancreatic cancer are widely recognized. Despite the development of several new treatment regimens for pancreatic cancer, little if any benefit has been appreciated, leaving this disease as one of the most significant unmet medical needs in cancer.

NPC-1C is a chimeric immunoglobulin molecule comprised from the variable region of the heavy chain and light chain of murine NPC-1, genetically engineered in-frame with the constant regions of a human IgG1 isotype. NPC-1, the predecessor of NPC-1C, was derived from a Tumor Associated Antigen (TAA) based vaccine that was previously tested in a Phase 1-2 clinical trial performed in the United States in the 1980's that explored the use of TAA therapy in patients with adenocarcinoma of the colon. These early studies demonstrated safety as well as preliminary evidence of activity in these patients treated with the vaccine.

NPC-1C antibody-staining studies demonstrate specific immunoreactivity with cancer tissues from colon and pancreas patients, whereas only weak binding, if at all, is observed in normal pancreas or colon tissues with no cross-reactivity observed in other normal human tissues. The Phase 2 portion of this trial is an open label, multi-center study estimated to treat approximately 30 patients with pancreatic cancer who have failed first line therapy, and 43 patients with metastatic colorectal cancer who are refractory to standard treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age: >/= 18
* Diagnosis:

  * Histologically confirmed recurrent, locally advanced unresectable or metastatic adenocarcinoma of the pancreas who have progressed after front line chemotherapy, OR
  * Histologically confirmed metastatic colorectal adenocarcinoma who have progressed after at least 2 standard chemotherapy regimens.
* Tumor sections must stain >/= 20% positive for NPC-1C antibody/antigen target
* Measurable disease (by RECIST)
* Karnofsky performance status of >/= 50%
* Laboratory Function (within 21 days of receiving first dose of study drug):

  * Hemoglobin > 8.5 g/dL, or on stable doses (hematocrit stable within 1 gram and dose stable for one month) of erythropoietin or similar medication.
  * Absolute neutrophil count (ANC) >/= 1,500/mm3
  * Platelets >/= 50,000/mm3
  * Total bilirubin </= 2.0 mg/dL
  * ALT and AST </= 2.5 times the ULN, or, if the patient has liver metastases, </= 5 times the ULN
  * Creatinine </= ULN
* Voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care.
* Expected to be able to remain on a study protocol for at least 8 weeks.
* Is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control for the duration of the study. Male subject agrees to use an acceptable barrier method for contraception during the study.

EXCLUSION CRITERIA:

* Has history of disseminated or uncontrolled brain metastases or central nervous system disease.
* Ascites with abdominal distention.
* Mechanical, non-reversible reason for not being able to eat, or have a likelihood of developing malignant bowel obstruction during the course of the induction phase of treatment; subjects with uncomplicated J-tubes will not be excluded.
* Any major surgery within four weeks of enrollment.
* Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Has another serious medical illness, including a second malignancy, or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Pregnant or breast-feeding.
* Any chemotherapeutic agents or corticosteroids within 2 weeks of study entry or biologic treatment within 4 weeks of study entry.
* Use of any high risk medications that prolong the QT/QTc interval.
* History of allergic reaction to Erbitux greater than grade 1.
* Uncontrolled diabetes.
* Prior history of a documented hemolytic event.
* Receiving warfarin.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by analysis of CT scans pre and post therapy, clinical laboratory tests, and physical examinations. | 10 weeks
Efficacy OS | 5 months
  Using the recommended phase 2 dose (RP2D) evaluate the overall survival (OS) associated with administration of NPC-1C (NEO-102) in subjects with metastatic, locally advanced unresectable or recurrent pancreatic cancer or metastatic colorectal cancer that express NPC-1C target on tumor.

SECONDARY OUTCOMES:
Safety will be assessed by analysis of adverse experiences, clinical laboratory tests, and physical examinations. | 10 weeks
Pharmacokinetics and select immune responses to the antibody will be assessed. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Arlen, M.D., Study Director — Precision Biologics, Inc
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas